CLINICAL TRIAL: NCT04688346
Title: Cardiovascular Effects of Racemic Epinephrine Pellets Used in Pediatric Restorative Dentistry Under General Anesthesia
Brief Title: Cardiovascular Effects of Racemic Epinephrine Pellets
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Travis Nelson, Clinical Associate Professor, School of Dentistry, University of Washington
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: STUDY00006670
Record Dates: First submitted 2020-11-02; First posted 2020-12-30 (Actual); Results first posted 2021-05-13 (Actual); Last update posted 2021-05-13 (Actual); Status verified 2021-05

CONDITIONS: Epinephrine Causing Adverse Effects in Therapeutic Use

STUDY DESIGN:
Intervention Model Description: This is a, single-blinded, placebo-controlled, split-mouth randomized trial. A sample size of 20 pediatric patients will be used for this pilot study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (Placebo Comparator): Saline Pellet
  Interventions: Drug: HemeRX epinephrine pellets
- Intervention (Experimental): Racemic Epinephrine Pellet
  Interventions: Drug: HemeRX epinephrine pellets

INTERVENTIONS:
Drug: HemeRX epinephrine pellets — Racemic Epinephrine Pellet

SUMMARY:
The primary aim of this study was to determine if topical racemic epinephrine pellets affect heart rate (HR), systolic blood pressure (SBP), diastolic blood pressure (DBP) or mean arterial pressure (MAP) in children receiving dental care under general anesthesia (GA). Thirteen patients requiring prefabricated zirconia crowns on both primary maxillary first molars were recruited into a split-mouth randomized controlled pilot study. Patients received a continuous infusion of propofol and remifentanil with inhaled nitrous oxide/oxygen. After patient randomization and tooth preparation, either saline pellets (control) or racemic epinephrine pellets (treatment) were applied directly to gingival tissue. Vital sign measurements were recorded for 5 minutes. The procedure was repeated with either control or treatment on the contralateral side.

DETAILED DESCRIPTION:
Dental caries is the most common chronic disease of childhood. 3-6% of US children experience early childhood caries, a condition that may necessitate restorative dental treatment. Prefabricated crowns are the treatment of choice for children with rampant caries involving large or multiple surface lesions or developmental defects. In such situations, crowns reinforce the tooth and provide increased durability and longevity over intracoronal restorations such as fillings. They also reduce the chance that the tooth will experience recurrent decay.

In routine clinical practice, preformed metal crowns, also known as stainless steel crowns (SSC) are frequently indicated due to their extreme durability, relatively low cost, and minimal technique sensitivity. Stainless steel crowns (SSC) are no longer the only standard of care in restoring primary teeth. Although SSCs are highly effective, esthetics can be a concern for parents. Prefabricated zirconia crowns provide an esthetic solution. Zirconia is a crystalline dioxide of zirconium that has mechanical properties similar to those of metals while its color is similar to that of teeth. According to a recent randomized controlled trial, both SSC and zirconia crowns proved to be an excellent choice for molar teeth full coverage restorations. However, zirconia crowns performed better from the standpoint of esthetics, gum tissue response and plaque retention. (Abdulhadi Bashaer S, Abdullah Medhat M, et al. Clinical evaluation between zirconia crowns and stainless steel crowns in primary molars teeth. Journal of pediatric dentistry. 2017, Vol 5, issue 1; 21-27.)

Both Stainless steel crown and zirconia crown preparations include removing caries, followed by reducing the height of the tooth by 1.5 mm, reducing the sides of the tooth to make the pre-fabricated crown fit on the tooth. The SSC preparation requires subgingival reduction 1-2 mm below the gumline on anterior and posterior surfaces (not medial and lateral). The only additional preparation step that zirconia crown preparation involves is medial and lateral reduction of the tooth; therefore, there is little additional time that is needed for preparation of the crown since the only difference is the depth of the side reduction and preparing it circumferentially. In addition, the Primary Investigator (PI) is the provider who will be treating all patients. The PI is an experienced pediatric dentist and has been providing both types of crowns to patients under general anesthesia every week for many years.

The average time for a dental procedure under general anesthesia is between 1-3 hours. Factors that increase time include extent of disease, number of fillings/crowns placed, and pediatric dentist's experience.

The pediatric dentist that will be doing the surgery on all patients has been practicing for many years and has prepared thousands of SSC and zirconia crowns. Therefore, it is not anticipated that it will require additional time to prepare the zirconia crowns versus stainless steel crowns.

Vital signs (BP and HR) will be monitored for 4 minutes/tooth, 5-8 minutes total (See attached chart showing the difference). During this time the patient will be continuously anesthetized and under close observation by the attending anesthesiologist. This constitutes a minimal risk to a child's health.

According to studies, epinephrine half-life is about two minutes and once the epinephrine pellet is removed, concentrations will drop by 93.75% over 4 half-lives which is about 8 minutes. Therefore, if there is any effect on blood pressure it will show immediately and will go back to normal within the time frame that we are recording data. The procedure will be stopped if the blood pressure is at a harmful range to patient.

All children will have both of their maxillary primary first molars (#B, #I) prepared for prefabricated Zirconia crowns. Teeth that require pulpotomy or pulpectomy treatment will be excluded from the study.

In the control group, hemostasis will be achieved by using two pellets soaked with 0.9% sodium chloride (physiological saline). In the intervention group, hemostasis will be achieved by using two racemic epinephrine HCl pellets (HemeRX, Racellet #3, Sprig Oral Health Technologies, Inc. Loomis, CA). Racellet #3 contains an average of 0.55 mg (0.42 to 0.68 mg/pellet) of racemic epinephrine hydrochloride per pellet.

A standard general anesthesia protocol will be used during the study. All monitoring equipment will be applied at this time for the measurement of vital signs throughout the anesthesia. Vital signs will include: respiratory rate, oxygen-saturated hemoglobin percentage, heart rate (HR) in beats per minute (bpm) and cardiac rhythm, which will be continuously recorded from a 3-lead electrocardiogram (ECG). The systolic blood pressures (SBP) and diastolic blood pressures (DBP) will be measured in millimeters of mercury (mmHg) via ankle artery cuff connected to monitors.

Investigators will use a randomization software before the enrollment of the first subject to randomly determine if the right or the left side of the mouth will be the intervention. Once consent is obtained, randomization software will be used again to determine whether the patient will be given control or intervention treatment first. Once patients are under anesthesia and after other dental treatments are completed, the maxillary first primary molars (#B, #I) will be prepared for Zirconia crowns. The crowns will be prepared independently. One tooth will be prepared first, the pre-fabricated crown will be tried on to make sure the fit is correct. Next either intervention or control pellets will be placed around the gumline of the tooth and removed after one minute. The vital signs will continue to be recorded for the next 4 minutes meanwhile he crown is being cemented on the tooth. Once that is done the operator will move to the other tooth and repeat the same steps.

The process of preparing the tooth for a Zirconia crown requires a circumferential subgingival preparation. Tissue irritation and bleeding is inherent in this process. Once the crown is ready to be permanently cemented hemostasis becomes very important. In both the control and intervention group of teeth, two pellets will be applied directly around the gingival tissue of the prepared tooth and held for one minute with direct pressure and then removed based on the manufacturer's recommendation. The time of application will be recorded. The adequacy of hemostasis will be determined subjectively by the attending dentist and recorded as "adequate" or "inadequate" at 1, 2, 3, 4, and 5 minutes after placement. Adequate hemostasis is defined as gingival tissue being dry and hemorrhage-free. Inadequate hemostasis is defined as inability to keep the gingival tissue dry and without hemorrhage. If hemostasis is not achieved after four minutes of managing a subject during the study intervention (saline or epinephrine pellets) to which a tooth has been randomized, we will revert to the standard of care in order to stop the bleeding. Lidocaine will not be administered as a primary local anesthetic nor would it be used during our study. Only epinephrine pellets and saline pellets will be used in the study for achieving hemostasis.

Cardiovascular outcomes of patient's systolic blood pressure (SBP), diastolic blood pressure (DBP) and heart rate (HR) will be collected by the graduate researcher during the procedure. The researcher will record the blood pressure/HR before placement of pellets, immediately after placement and at 1, 2, 3, 4, 5 minutes after placement. The pellets will stay on the tissue for 1 minute only and then removed. The researcher will also record hemostasis efficacy as per dental surgeon as either "adequate" or "inadequate" during the procedure.

In addition to the above measurements, cardiac rhythms will be assessed continuously via ECG and recording any arrhythmias. Mean arterial pressure (MAP), the amount of time in surgery and anesthesia medications used for each patient will also be recorded. All patients will be discharged on the same day after adequate recovery observation time.

ELIGIBILITY:
Inclusion Criteria:

1. Children ages 2-9 years undergoing general anesthesia for comprehensive dental treatment at the University of Washington Center of Pediatric Dentistry.
2. Healthy patients according to the American Society of Anesthesiologists (ASA) classification I or II.
3. Patients who have caries lesions requiring prefabricated crowns on primary maxillary first molars #B and #I.

Exclusion Criteria:

1. Pediatric patients with any severe systemic illness (ASA Classification III or greater).
2. Pediatric patients with known cardiac arrhythmia, cardiovascular disease, diabetes and thyroid disease.
3. Patients who are taking anti-arrhythmic, antihypertensive, or ionotropic medications.
4. Patients who would need pulpotomy or pulpectomy treatment on primary maxillary first molars #B and I.

Ages: 2 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 13 (Actual)
Dates: Start 2019-06-10 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2019-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Travis M Nelson, DDS, Principal Investigator — University of Washington
Locations (1):
- UW Center for Pediatric Dentistry, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 13 participants were enrolled. Each served as their own control. Left side primary maxillary molar received Saline, right side received Epinephrine pellets.
Units Other Than Participants: Primary Maxillary Molar Teeth
Groups:
- Saline First, Then Epinephrine: Saline Pellet
  HemeRX epinephrine pellets: Racemic Epinephrine Pellet
- First Epinephrine, Then Saline: Racemic Epinephrine Pellet
  HemeRX epinephrine pellets: Racemic Epinephrine Pellet
Period: Overall Study
Arm/Group | Saline First, Then Epinephrine | First Epinephrine, Then Saline
Started | 6; 6 Primary Maxillary Molar Teeth | 7; 7 Primary Maxillary Molar Teeth
First Intervention | 6; 6 Primary Maxillary Molar Teeth | 7; 7 Primary Maxillary Molar Teeth
Second Intervention | 6; 6 Primary Maxillary Molar Teeth | 7; 7 Primary Maxillary Molar Teeth
Completed | 6; 6 Primary Maxillary Molar Teeth | 7; 7 Primary Maxillary Molar Teeth
Not Completed | 0; 0 Primary Maxillary Molar Teeth | 0; 0 Primary Maxillary Molar Teeth

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Saline First, Then Epinephrine | First Epinephrine, Then Saline | Total
Number analyzed (Participants) | 6 | 7 | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 4.9 (1.5) | 4.5 (1.7) | 4.7 (1.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 3 | 4 | 7
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 6 | 7 | 13

OUTCOME MEASURES:

1. Primary Outcome: Cardiovascular Outcomes
Description: To determine heart rate change of patients receiving treatment with topical racemic epinephrine compared to those receiving a placebo.
Time Frame: 5 minutes
Measure: Mean (Standard Deviation); unit: Beats Per Minute
Arm/Group | Control | Intervention
Number analyzed (Participants) | 13 | 13
Beats Per Minute | 91.5 (18.2) | 93.4 (15.1)

2. Primary Outcome: Cardiovascular Outcomes
Description: To determine blood pressure change of patients receiving treatment with topical racemic epinephrine compared to those receiving a placebo.
Time Frame: 5 minutes
Measure: Mean (Standard Deviation); unit: mmhg
Arm/Group | Control | Intervention
Number analyzed (Participants) | 13 | 13
mmhg | -3.1 (5.1) | -2.7 (3.6)

3. Secondary Outcome: Hemostasis Efficacy
Description: To determine time to achieving hemostasis (based upon subjective assessment of surgeon) on patients receiving treatment with topical racemic epinephrine compared to those receiving a placebo.
Time Frame: 5 minutes
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Control | Intervention
Number analyzed (Participants) | 13 | 13
Minutes | 4.2 (2) | 2.2 (2)
Statistical Analysis 1: Comparison: Control vs Intervention; Test type: Non-Inferiority — t-test; p = 0.05, t-test, 2 sided; Mean Difference (Final Values) = 1

ADVERSE EVENTS:
Time Frame: Participants were assessed for adverse outcomes during the period of their general anesthesia visit (1 day).
Description: cardiac and hematological adverse outcomes
Arm/Group | Control | Intervention
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/13
Other Adverse Events (participants affected / at risk) | 0/13 | 0/13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-12-23): https://cdn.clinicaltrials.gov/large-docs/46/NCT04688346/Prot_SAP_000.pdf